CLINICAL TRIAL: NCT00295191
Title: Multiple Interventions Related to Dialysis Procedures in Order to Reduce Cardiovascular Morbidity and Mortality in Hemodialysis Patients: Prospective, Randomized, Controlled Study
Brief Title: Multiple Interventions Related to Dialysis Procedures in Order to Reduce Cardiovascular Morbidity and Mortality in HD Patients(EGESTUDY)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Principal Investigator, Ercan OK, Principal Investigator, Ege University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EGE99803466003
Record Dates: First submitted 2006-02-22; First posted 2006-02-23 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: End-stage Renal Disease; Hemodialysis
Keywords: end-stage renal disease; hemodialysis; cardiovascular morbidity and mortality; high flux dialyser; ultrapure dialysate; coronary vascular calcifications; carotid intima-media thickness; atherosclerosis
MeSH Terms: conditions — Kidney Failure, Chronic; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): high-flux dialyser
  Interventions: Procedure: high-flux membrane
- 2 (Active Comparator): low-flux dialyser
  Interventions: Procedure: low-flux membrane
- 3 (Active Comparator): conventional dialysate
  Interventions: Procedure: conventional dialysate
- 4 (Active Comparator): ultrapure dialysate
  Interventions: Procedure: ultrapure dialysate

INTERVENTIONS:
Procedure: high-flux membrane — high-flux dialyser
  Arms: 1
Procedure: low-flux membrane — low-flux dialyser
  Arms: 2
Procedure: conventional dialysate — conventional dialysate
  Arms: 3
Procedure: ultrapure dialysate — ultrapure dialysate
  Arms: 4

SUMMARY:
This study aims to investigate the effects of high flux dialyser use and ultra pure dialysate utilization on cardiovascular disease by evaluating cardiovascular morbidity and mortality, progression of carotid artery intima-media thickness and coronary artery calcifications, inflammatory state, lipid levels, nutritional status, and erythropoietin requirement in hemodialysis patient population. It is hypothesized that both interventions in this project may diminish cardiovascular disease in hemodialysis patients.

DETAILED DESCRIPTION:
This proposed prospective, randomized, controlled study aims to investigate the effects of high flux dialyser use and ultra pure dialysate utilization on cardiovascular disease by evaluating cardiovascular morbidity and mortality, progression of carotid artery intima-media thickness and coronary artery calcifications, inflammatory state, lipid levels, nutritional status, and erythropoietin requirement in hemodialysis patient population. It is hypothesized that both interventions in this project may diminish cardiovascular disease in hemodialysis patients.

Their beneficial effects may be directly represented by significantly reduced cardiovascular morbidity and mortality. The proposed additional investigations, such as a possible decrease in the progression of coronary artery calcification and carotid artery intima-media thickness, will help us to understand the mechanisms of the expected reduction or serve as surrogate markers of atherosclerosis, in case the benefit of the interventions cannot be proven with statistical significance.

Seven hundred and four hemodialysis patients treated in Ege University Hospital Dialysis Unit and eight FMC Clinics will be enrolled into the study (3-year follow-up; percentage of yearly expected end-point 10%;expected event-free survival rate for control group during three year is 72.9%,a bilateral alpha risk equal to 5%; an 90% power to detect an increase of 15% in event-free survival at the end of 3-year follow-up in favor of the each intervention group). Annual drop-out rate is estimated as %15-20.

It is designed as 2x2 factorial; the cases, first, will be randomized to high flux dialyser and low flux dialyser arms; then, they will be re-randomized to ultra pure (online-produced by using Diasafe and checked by endotoxin measurement) and standard dialysate arms. The study will last three years; an intermediate analysis will be performed at the 18th month.

Primary end-point is the composite of cardiovascular mortality and myocardial infarction, stroke, revascularization, unstable angina pectoris requiring hospitalization (at 18 ad 36th month).

Secondary end-points are overall mortality, progression of coronary artery calcification, progression of carotid artery intima-media thickness, changes in post-dialysis body weight and upper mid-arm circumference, hematocrit and related rHu-EPO doses, changes in the levels of albumin, transferrin, total cholesterol, triglyceride, HDL cholesterol, LDL cholesterol, high sensitive CRP, and β-2 microglobulin.

At the 0-18-36 months, coronary artery calcification will be assessed by multi-slice CT and carotid artery intima-media thickness by B-mode ultrasonography. Lipids and CRP will be measured in every three months.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years
* On maintenance bicarbonate hemodialysis scheduled thrice weekly, at least 12 hours/week
* Willingness to participate in the study with a written informed consent.

Exclusion Criteria:

* To be scheduled for living donor renal transplantation
* To have serious life-limiting co-morbid situations; namely active malignancy, active infection, end-stage cardiac, pulmonary, or hepatic disease; pregnancy or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2005-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
cardiovascular mortality, myocardial infarction, stroke, unstable angina pectoris requiring hospitalization, revascularization | three years

SECONDARY OUTCOMES:
overall mortality | three years
progression of coronary artery calcification | three years
progression of carotid artery intima-media thickness | three years
changes in post-dialysis body weight | three years
changes in upper mid-arm circumference | three years
changes in hematocrit and related rHu-EPO doses | three years
changes in the levels of albumin, transferrin, total cholesterol, triglyceride, HDL cholesterol, LDL cholesterol, high sensitive CRP, and β-2 microglobulin. | three years

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Ok, M.D, Principal Investigator — Ege University School of Medicine Nephrology Department
Locations (2):
- Turkey (Türkiye) (2):
  - FMC Clinics, Bornova, İzmir
  - Ege University School of Medicine, Bornova-Izmir

REFERENCES:
- [Derived] Ok ES, Asci G, Toz H, Ritz E, Kircelli F, Sever MS, Ozkahya M, Sipahi S, Dheir H, Bozkurt D, Omer Z, Sahin OZ, Ertilav M, Ok E. Glycated hemoglobin predicts overall and cardiovascular mortality in non-diabetic hemodialysis patients. Clin Nephrol. 2014 Sep;82(3):173-80. doi: 10.5414/cn108251. PMID 25079862